CLINICAL TRIAL: NCT07294014
Title: Investigation of Medial Longitudinal Arch and Foot Function in Patients With Lipedema: A Cross-Sectional Study
Brief Title: Investigation of Medial Longitudinal Arch and Foot Function in Patients With Lipedema
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: Marmara-FTR-GNY-02
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lipedema; Hypermobility Syndrome (Disorder); Pes Planus; Joint Hypermobility
Keywords: lipedema; mypermobility; foot function; pes planus; joint hyper mobility; foot morphology; Meary angle; calcaneal inclination angle
MeSH Terms: conditions — Lipedema; Flatfoot; Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lipedema group: Participants diagnosed with lipedema based on established clinical criteria, including characteristic bilateral lower-extremity adipose tissue enlargement, pain or tenderness on palpation, easy bruising, and preservation of foot anatomy. Diagnosis is confirmed by a physiatrist or relevant specialist through medical history and physical examination. These participants will undergo radiographic foot assessment, hypermobility evaluation, and functional testing as part of the study protocol.
- Control group: Age- and BMI-matched female participants presenting with nonspecific foot pain but without a diagnosis or clinical suspicion of lipedema, lymphedema, connective tissue disorders, or systemic inflammatory disease. These individuals will undergo the same radiographic, hypermobility, and functional assessments as the lipedema group, allowing for direct comparison of foot morphology and joint mobility parameters.

SUMMARY:
Lipedema is a chronic adipose tissue disorder that commonly leads to joint laxity, hypermobility, and functional limitations, yet its impact on foot morphology has not been systematically examined. This case-control study aims to investigate whether patients with lipedema exhibit a higher prevalence of generalized joint hypermobility and foot structural abnormalities-specifically pes planus-compared with age- and BMI-matched controls. Using radiographic measurements (Meary angle and calcaneal inclination angle), clinical hypermobility assessment, and validated functional scales, the study seeks to determine the relationship between lipedema, hypermobility, and foot function.

DETAILED DESCRIPTION:
Lipedema is a progressive adipose tissue disorder characterized by disproportionate subcutaneous fat accumulation, predominantly in the lower extremities. Patients frequently experience pain, easy bruising, reduced quality of life, and musculoskeletal complications such as joint laxity and hypermobility. Although previous studies have suggested an increased prevalence of hypermobility in individuals with lipedema, the potential impact of these biomechanical changes on foot posture and foot function remains insufficiently studied.

This case-control, single-session, single-blind (participant-blinded) study is designed to evaluate structural and functional foot characteristics in women diagnosed with lipedema, compared with age- and BMI-matched controls presenting with nonspecific foot pain. The primary radiographic variables include the Meary angle and calcaneal inclination angle measured on standardized lateral foot radiographs. These measurements provide objective quantification of midfoot alignment and arch height, enabling detection of pes planus and related morphological deviations.

In addition to radiographic assessment, the study incorporates established clinical tools to quantify joint hypermobility, foot function, pain severity, and physical activity levels. The Beighton score will be used to determine generalized joint hypermobility. Functional and symptomatic status will be evaluated using validated questionnaires, including the Foot Function Index (FFI), Lower Extremity Functional Scale (LEFS), Visual Analog Scale (VAS) for pain, and the International Physical Activity Questionnaire-Short Form (IPAQ-SF).

Sociodemographic and clinical data-including disease duration, comorbidities, and lower extremity volumetric measurements-will be systematically recorded to identify potential associations between patient characteristics and foot morphology. The study aims to clarify whether the presence of hypermobility in lipedema contributes to alterations in medial longitudinal arch structure and whether these changes are more prevalent than in a matched control population.

The findings are expected to provide insight into the biomechanical consequences of lipedema, support more accurate clinical assessment, and potentially guide rehabilitative strategies targeting lower extremity alignment and function in this patient group.

ELIGIBILITY:
General Inclusion Criteria (Apply to All Participants)

* Female participants
* Age 18 years or older
* Able to read and write (literacy requirement)
* Availability of bilateral lateral foot radiographs obtained within the past 1 year in the hospital PACS system
* Willing and able to provide written and verbal informed consent

Additional eligibility criteria for Lipedema Group

- Clinical diagnosis of lipedema according to Halk and Damstra criteria.

Additional eligibility criteria for Control group:

* Female patients presenting with nonspecific foot pain
* Similar age and BMI range as the lipedema group
* No clinical diagnosis or suspicion of lipedema

Exclusion Criteria (Apply to all participants)

* Pregnancy
* Illiteracy
* Inability or unwillingness to provide written and verbal informed consent
* History of lower extremity fracture, trauma, or orthopedic surgery
* Diagnosis of diabetes mellitus
* Known rheumatologic disease
* Known polyneuropathy or peripheral nerve injury affecting the lower extremities

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients presenting to the Physical Medicine and Rehabilitation outpatient clinics at Marmara University Pendik Training and Research Hospital will be screened for eligibility. The study population will include women clinically diagnosed with lipedema according to established diagnostic criteria, as well as age- and BMI-matched female patients with nonspecific foot pain who will serve as the control group.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Meary angle (Degrees) | Day 1
  The Meary angle (talo-first metatarsal angle) will be measured on standardized lateral foot radiographs to evaluate medial longitudinal arch alignment. Increased angles indicate midfoot collapse and are used to identify pes planus. Higher values represent greater deviation from normal alignment.
Calcaneal Inclination Angle (Degrees) | Day 1
  The calcaneal inclination angle will be measured on lateral foot radiographs to assess arch height. Lower angles indicate reduced arch height, consistent with pes planus. Measurements are obtained using established radiographic guidelines.

SECONDARY OUTCOMES:
Beighton Score (0-9) | Day 1
  Generalized joint hypermobility will be evaluated using the Beighton Score, a validated 9-point scale assessing joint laxity in the fingers, elbows, knees, and spine. A score ≥4 indicates generalized hypermobility.
Lower Extremity Functional Scale (LEFS) Score | Day 1
  The LEFS questionnaire assesses lower-extremity functional status across daily activities. Scores range from 0 to 80, with higher scores indicating better function.
Foot Function Index (FFI) Total Score | Day 1
  The FFI evaluates foot-related disability and pain using 23 items across three subscales: pain, disability, and activity limitation. Higher scores reflect greater functional impairment.
Visual Analog Scale (VAS) for Pain (0-100 mm) | Day 1
  Pain severity in both lower extremities will be assessed in three conditions:
  VAS-Movement VAS-Rest VAS-Night Higher values indicate greater pain intensity.
Physical Activity Level (IPAQ-Short Form) | Day 1
  Physical activity levels will be assessed using the International Physical Activity Questionnaire-Short Form. Results will classify participants into low, moderate, or high activity categories based on metabolic equivalent (MET)-minutes per week.

OTHER OUTCOMES:
Lower Extremity Volumetric Measurements (cm or mL) - Lipedema Group Only | Day 1
  Circumferential measurements at standardized anatomical points will be used to calculate volumetric estimates of lower extremity adipose tissue distribution to support characterization of disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available 6 months after publication of the main results and remain accessible for at least 5 years following publication.
Access Criteria: Qualified researchers may request access to the de-identified dataset and supporting documentation by submitting a brief research proposal and data access agreement to the corresponding investigator (Gökçenur Yalçın, M.D., Department of Physical Medicine and Rehabilitation, Marmara University, Istanbul, Turkey). Data will be shared via a secure institutional data repository upon approval by the principal investigator and the Marmara University Ethics Committee.